CLINICAL TRIAL: NCT06303076
Title: Efficacy of Tizanidine (0.1 mg/Kg/HS) Versus Zolpidem 10 mg HS in Primary Insomnia: Double Blind Randomized Controlled Trial
Brief Title: Tizanidine vs. Zolpidem in Primary Insomnia: A Randomized Trial
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Sultan Qaboos University (Other)
Responsible Party: Principal Investigator, Mohammed Al Alawi, Dr Mohmmed Al Alawi Bsc, MD,PhD, MRCPsych, OMSBPsych, ARABPsych, Sultan Qaboos University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 134
Record Dates: First submitted 2024-03-04; First posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Depressive Disorder, Major
MeSH Terms: conditions — Depressive Disorder, Major | interventions — tizanidine; Zolpidem

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tizanidine Group (Experimental): Participants will be asked to ingest Tinazidine, orally at home immediately before going to bed to sleep. Initially, the patients will be asked to ingest 2 mg HS, and it will be titrated up by 2 mg every 4 days, as per response and tolerability, up to a maximum dose of 0.1 mg/kg/HS.
  Interventions: Drug: Tizanidine Hcl 4Mg Tab
- Zolpidem Group (Active Comparator): Participants will be asked to ingest Zolpidem 10 mg HS, orally at home before bedtime.
  Interventions: Drug: Zolpidem Tartrate 10 mg

INTERVENTIONS:
Drug: Tizanidine Hcl 4Mg Tab — Initial Dose Administration:
  Patients will start by taking an initial dose of 2 mg of Tizanidine at bedtime (HS).
  Dose Titration Process:
  Every 4 days, the dose of Tizanidine will be increased by 2 mg. This titration is based on the patient's response to the medication and their tolerability of it.
  Maximum Dose Limit:
  The dose titration will continue until reaching the maximum dose of 0.1 mg/kg/HS, or until the maximum tolerated dose is identified, whichever comes first.
  Monitoring and Adjustment:
  Throughout the titration process, patients will be closely monitored for any adverse effects and for the effectiveness of the medication.
  Adjustments to the dosing schedule may be made based on the clinician's assessment of tolerability and therapeutic response.
  Arms: Tizanidine Group
Drug: Zolpidem Tartrate 10 mg — nitial Dose Administration:
  Participants will start by taking an initial dose of Zolpidem 5 mg orally at home before bedtime (HS).
  Response Evaluation and Dose Adjustment:
  If there is no response to the initial 5 mg dose and it is tolerated well by the participant, the dose will be increased to 10 mg.
  Monitoring and Adjustment:
  Participants will be monitored for their response to the medication as well as for any adverse effects.
  The decision to increase the dose to 10 mg will be based on the absence of a therapeutic response to the initial dose and the participant's tolerability of Zolpidem.
  Dose Maximization and Safety:
  The increase to a 10 mg dose is aimed at maximizing therapeutic efficacy while ensuring the safety and tolerability of the medication in participants who do not respond to the lower dose.
  Arms: Zolpidem Group

SUMMARY:
The study's primary objective is to evaluate the effectiveness of Tinazidine compared to Zolpidem in enhancing sleep quality, with secondary objectives including the assessment of adverse effects, safety profile, and patient tolerance with each treatment. The trial will be conducted as a double-blind RCT, with participants randomly assigned to receive either Tinazidine (0.1 mg/Kg/HS) or Zolpidem 10 mg HS, for 12 weeks. Eligible participants, aged 18-60 years, diagnosed with primary insomnia as per DSM-5 criteria, will be recruited from an outpatient sleep clinic affiliated with Al-Masara Hospital. Data on sleep quality, and side effects, will be collected using the Sleep Pittsburgh Sleep Quality Index (PSQI), Clinical Global Impression (CGI), sleep diaries, actigraphy, polysomnography, and regular clinical interview though OPD follow-up visits. The primary outcome considered was the mean global PSQI score before and after the treatment. The primary outcome will be measured four times (baseline, 4 weeks, 8 weeks, and 12 weeks), We considered an attrition rate (dropout/lost follow-up) of 10%. Therefore, the sample size is 90 subjects (45 in each group). Group comparisons for mean scores will be conducted using independent samples t-tests, and within-group comparisons will be assessed using paired samples t-tests. Changes in sleep quality over time between treatment groups will be evaluated using repeated measures ANOVA. Associations between categorical variables will be examined using Chi-square tests (including Fisher's exact or Likelihood ratio tests as appropriate). Statistical significance will be considered for p-values less than 0.05. All analyses will be performed using IBM SPSS Statistics (Version 29.0). The findings of this study seek to elucidate the comparative efficacy and safety profiles of Tizanidine and Zolpidem in treating primary insomnia. The study aims to offer insights into the effectiveness of Tizanidine versus Zolpidem in improving sleep quality among patients with primary insomnia. Through the evaluation of efficacy, adverse effects, and safety profiles. This study aims to inform clinicians and healthcare practitioners about the optimal treatment choices for individuals with primary insomnia.

DETAILED DESCRIPTION:
Efficacy of Tizanidine (0.1 mg/Kg/HS) versus Zolpidem 10 mg HS in Primary Insomnia: Double Blind Randomized Controlled Trial

Literature review:

Insomnia: Prevalence and Impact

Around 10% of adults have an insomnia disorder, while another 20% experience occasional insomnia symptoms (1). Women, older adults, and those facing socioeconomic challenges are more prone to insomnia. Insomnia often persists over time, with a 40% persistence rate over five years (1). Insomnia is a significant public health concern requiring individual clinical care and broad population-level interventions to improve sleep health (1).

The Individual and Public Health Ramifications of Insomnia

On an individual level, insomnia has significant repercussions on daily life, including impaired daytime function, emotional distress, reduced productivity, increased healthcare utilization, and heightened accident risk (2). Along with physiological hyperarousal, cardiometabolic morbidities such as hypertension, and diabetes, neurocognitive impairment such as short-term memory impairment, and psychological impairment such as depression, and anxiety (2)(3). Additionally, untreated insomnia tends not to improve over time (3).

On a public level, insomnia impacts various aspects of society. It contributes to an increased economic burden through decreased work productivity and higher healthcare costs due to increased healthcare service utilization (4). Additionally, insomnia heightens the risk of accidents, including traffic accidents, jeopardizing public safety (4). Its association with mental health disorders adds to the healthcare burden of managing these conditions, while the increased risk of chronic medical diseases further strains healthcare systems (5). Given that the untreated economic costs of insomnia far exceed that of treated insomnia (4), efforts should be focused on developing clinical trials aimed at assessing the cost-benefit, and cost-effectiveness of various insomnia therapies.

Defining Primary Insomnia According to DSM-5 Criteria

Primary insomnia, as defined in the DSM-5 criteria (6), refers to a sleep disorder characterized by difficulty initiating or maintaining sleep, or experiencing non-restorative sleep, for at least one month. Individuals with primary insomnia often report significant distress or impairment in social, occupational, or other important areas of functioning due to their sleep difficulties. The DSM-5 criteria further specify that insomnia is not better explained by another sleep disorder, such as narcolepsy, or circadian rhythm sleep disorder, etc., and not due to another mental disorder. Additionally, the diagnosis of primary insomnia requires that the sleep disturbance does not occur due to the physiological effect of a medical condition or substance use (6).

Current FDA-Approved Medications for Insomnia

Current FDA-approved medications for insomnia include benzodiazepines, such as Triazolam, and Temazepam, as well as non-benzodiazepines (Z drug) such as zolpidem, and zaleplon. Additionally, melatonin agonist ramelteon, tricyclic antidepressant doxepin, and orexin antagonists such as suvorexant are also among the approved options for managing insomnia (7).

Zolpidem was the first Z drug to be developed. In studies investigating zolpidem adverse events that arose during treatment, such as drowsiness, nausea, dizziness, nightmares, and agitation, have led to the discontinuation of the zolpidem (7). Additionally, some patients experienced anterograde amnesia (7). Moreover, concerns about the frequent use of benzodiazepine for insomnia include the risk of dependence, drug-seeking behavior, and abuse in the context of inadequate medical supervision (8). Evaluating any new pharmacological treatments against conventional benzodiazepine and z-drugs intake is crucial, as there is limited data on the benefit-to-risk ratio of such treatment strategies, necessitating head-to-head trials.

Therapeutic Applications of Tizanidine

Tizanidine, a centrally acting alpha-2 agonist, is commonly prescribed to manage spasticity induced by conditions such as multiple sclerosis, stroke, and spinal cord injury. Beyond its labeled indications, it finds off-label use in alleviating chronic neck and back pain as well as chronic migraines (9).

Clinical Trials of Tizanidine in the Context of Insomnia

Tizanidine has shown promise in previous studies for its efficacy in sleep disturbances. In a study where 24 subjects with Myofascial pain syndrome received tizanidine, which was titrated up to 12 mg over 3 weeks and maintained for 2 weeks. the study results showed Pain intensity and disability decreased significantly from baseline at weeks 3 and 5 and after washout (P < .001). Pressure threshold and sleep improved for all study periods (P < .001). The Sleep in this study was assessed via a visual analog scale (VAS) (10).

In a randomized controlled clinical trial assessing the efficacy of adding either tizanidine or cyclobenzaprine in treating jaw pain, 45 patients diagnosed with myofascial pain were randomly assigned to three groups: a placebo group, a tizanidine group (4 mg), and a cyclobenzaprine group (10 mg). Patients were assessed for changes in pain intensity using the modified Severity Symptoms Index and changes in sleep quality using the Pittsburgh Sleep Quality Index. Results showed that all three groups experienced a reduction in pain symptoms and an improvement in sleep quality when comparing pretreatment and treatment scores (11).

An open-label dose-titration study investigated the effectiveness and tolerability of tizanidine hydrochloride tablets in preventing chronic daily headaches. The dosage was gradually increased from 2 mg at bedtime to a median daily dose of 14 mg (mean 13.5; SD 4.3; range 4 to 20), divided over three doses per day by the fourth week of treatment. Significant improvements were observed in overall headache status, mood, sleep, quality of life (P < .00001), as well as sexual function (P = .0075), and the Beck Depression Inventory-II scores (P = .00073). Mild-to-moderate adverse events reported by 10% of patients included somnolence, asthenia, and dry mouth. Three patients discontinued treatment due to somnolence, dry mouth, or constipation. Additionally, one patient experienced elevated liver enzymes which normalized after discontinuing the medication (12).

Adverse Effects and Pharmacokinetic Considerations of Tizanidine

Adverse reactions associated with tizanidine include hypotension, bradycardia, or excessive sedation requiring gradual dose reduction or stopping therapy (9). Given its extensive hepatic metabolism, tizanidine's pharmacokinetics can be significantly altered in patients with hepatic impairment. Thus, special attention must be given to the dosing and monitoring of tizanidine in such individuals to mitigate risks (9). Similarly, patients with renal impairment, particularly those with a creatinine clearance below 25 mL/min, require careful management when using tizanidine. Initiation at lower doses, along with close monitoring of therapeutic response, is recommended (9). Any decision to prescribe tizanidine during pregnancy should involve a thorough risk-benefit assessment to ensure the safety of both the mother and the fetus. Moreover, considering tizanidine's lipid-soluble nature, potential transfer into breast milk raises concerns regarding its use during lactation (9). Smoking has been identified as a factor that reduces tizanidine's plasma concentration and exposure, as observed in studies such as Al-Ghazawi et al. (13)

Following oral administration of tizanidine, the peak plasma concentrations occurred 1 hour after with a half-life of approximately 2 hours. (14). The doses employed in the present study constitute an initial dose of 2 mg HS, and it will be titrated up by 2 mg every 4 days, as per response and tolerability, up to a maximum dose of 0.1 mg/kg/HS administered before bedtime. This proposed dose was found effective in a clinical trial assessing the effects of tizanidine for refractory sleep disturbance in disabled children with spastic quadriplegia. The clinical trial included 21 children diagnosed with spastic quadriplegia and experiencing severe sleep disturbances. All these children exhibited abnormalities in both falling asleep and staying asleep. Tizanidine was administered at a dosage ranging from 0.1 to 0.2 mg/kg/day, divided into two or three doses. If daytime drowsiness was significant, tizanidine administration was limited to just before bedtime. Improvement in sleep induction and/or maintenance was observed in 13 patients (61.9%). Moreover, the families of the patients expressed satisfaction with the treatment (15).

The objective of this study was to compare in a double-blind design the subjective hypnotic efficacy and safety of Tizanidine (0.1 mg/kg/day), and a Zolpidem 10 mg HS over 12 weeks in adult patients with primary insomnia.

Study Objectives

Primary Objective:

To evaluate the efficacy of Tizanidine compared to Zolpidem in improving sleep quality among patients with primary insomnia.

Secondary Objectives:

* To assess the safety and side effect profile of Tizanidine.
* To compare patient tolerance and satisfaction between Tizanidine and Zolpidem treatments.

Hypotheses

Main Hypothesis:

Tizanidine is effective in the treatment of primary insomnia, offering a better safety profile with fewer side effects.

Secondary Hypotheses:

* Patients treated with Tizanidine will report fewer side effects compared to those treated with Zolpidem.
* Tizanidine will demonstrate higher patient tolerance and satisfaction in the treatment of primary insomnia.

Methodology

Study Design:

This study will be conducted as a double-blind, randomized controlled trial. Participants will be randomly assigned to receive either Tizanidine or Zolpidem for 12 weeks.

The trial design is a parallel-group randomized controlled trial. Participants will be randomly assigned to either one of the two treatment groups: the Tizanidine group or the Zolpidem group. This design allows for the comparison of the efficacy and safety of Tizanidine versus Zolpidem in the treatment of primary insomnia. The allocation ratio will be 1:1, ensuring an equal distribution of participants between the two treatment arms.

Trial setting:

The data were collected at the outpatient sleep clinic affiliated with Al-Masarah Hospital, Muscat, Oman.

Randomization:

The method used to generate the random allocation sequence:

The random allocation sequence was generated using a computerized random number generator.

The type of randomization:

Simple randomization was employed, where each participant had an equal chance of being assigned to either the tizanidine group or the Zolpidem group.

Study procedures:

Study medications:

* Tizanidine Group:

  * At all evenings and mornings during the treatment period at home, participants will be asked to document the sleep diaries and to wear the actigraphy. Sleep diaries are collected by the research assistant every week.
  * Every 4 weeks the patients will be asked to complete the questionnaires (Pittsburgh Sleep Quality Index (PSQI), and another self-report of suspected adverse drug reaction form).
  * At baseline, then in the 6th week, and 12th week of the treatment, the participants will be asked to attend the OPD for a clinical assessment by a specialist psychiatrist researcher. The Clinical Global Impression (CGI) scale (severity of illness, global improvement, and efficacy index) assessed by the researcher
  * Throughout the study, compliance was monitored by the research assistant calling the patients every other day in the morning.
  * Safety was assessed by adverse events (spontaneously reported by participants to the research assistant and/or assessed/observed by the researcher during the clinical follow-up visit in 6th week, and 12th week of the study) and vital signs (heart rate and blood pressure) at baseline, in 6th week, and 12th week of the treatment.
  * Polysomnography (PSG) at baseline and within one week of the end of the trial will be carried out.
  * At the end of the study period, a medical checkup by a medical officer will be carried out. In the medical check-up, a medical history will be carried out, a physical examination (including ECG) and laboratory evaluation will be performed within 1 week of the end of the study treatment.
* Zolpidem Group:

  * At all evenings and mornings during the treatment period at home, participants will be asked to document the sleep diaries and to wear the actigraphy.
  * Every 4 weeks the patients will be asked to complete the questionnaires (Pittsburgh Sleep Quality Index (PSQI), and another self-report of suspected adverse drug reaction form).
  * At baseline, then in the 6th week, and 12th week of the treatment, the participants will be asked to attend the OPD for a clinical assessment by a specialist psychiatrist researcher. The Clinical Global Impression (CGI) scale (severity of illness, global improvement, and efficacy index) assessed by the researcher
  * Throughout the study, compliance was monitored by the research assistant calling the patients every other day in the morning.
  * Safety was assessed by adverse events (spontaneously reported by participants to the research assistant and/or assessed/observed by the researcher during the clinical follow-up visit in 6th week, and 12th week of the study) and vital signs (heart rate and blood pressure) at baseline, in 6th week, and 12th week of the treatment.
  * Polysomnography (PSG) at baseline and within one week of the end of the trial will be carried out.
  * At the end of the study period, a medical checkup by a medical officer will be carried out. In the medical check-up, a medical history will be carried out, a physical examination (including ECG) and laboratory evaluation will be performed within 1 week of the end of the study treatment.
* Administration: Both medications will be administered orally, 30 minutes before bedtime.

Outcome Measures:

1. - Primary Outcome: Improvement in sleep quality, measured using the Pittsburgh Sleep Quality Index (PSQI).
2. - Secondary Outcomes: Frequency and severity of side effects, and patient satisfaction (assessed through a self-report of suspected adverse drug reaction form).

Data Collection Methods:

* Sleep diaries and actigraphy will be used to collect data on sleep patterns every morning, and every night.
* Standardized questionnaires at the 4th week, 8th week, and 12th week of the study include the Pittsburgh Sleep Quality Index (PSQI), and a self-report of suspected adverse drug reaction form.
* Clinical follow-up visits during the 4th week of intervention, 8th week of intervention, and the 12th week of intervention will be scheduled to monitor progress and gather subjective assessments.
* Polysomnography (PSG) at baseline and within one week of the end of the trial will be carried out.

Actigraphy

This is a method used to monitor activity and sleep-wake patterns over the study period. It involves wearing a small, wrist-worn device called an actigraph, which contains sensors that detect movement and record activity levels continuously.

Sleep diaries

These are self-reported records in which participants will be asked to track various aspects of their sleep-wake patterns over the study period. individuals are typically asked to fill out sleep diaries first thing in the morning, immediately upon waking up. The diaries will involve recording information about bedtime, wake-up time, sleep onset latency (time taken to fall asleep), wake after sleep onset (time spent awake during the sleep period), and any nighttime awakenings.

Polysomnography (PSG)

Polysomnography, a diagnostic examination employed during sleep, gathers physiological data through various sensors including electroencephalogram (EEG), electrooculogram (EOG), electromyogram (EMG), electrocardiogram (ECG), pulse oximetry, airflow, and respiratory effort.

Pittsburgh Sleep Quality Index (PSQI)

The Pittsburgh Sleep Quality Index (PSQI) is a self-administered questionnaire designed to evaluate sleep quality within one month. It comprises 19 specific items organized into seven components, ultimately generating a single global score. It is a widely used and validated instrument for assessing sleep quality in research and clinical settings. It has been extensively validated in various populations and has demonstrated good psychometric properties (17), including reliability and validity in the Arabic version (18). This scale is copyrighted and is owned by the University of Pittsburgh and may be reprinted & used without charge only for non-commercial research and educational purposes.

Clinical Global Impression

Self-report of suspected adverse drug reaction form

Patients will be asked to fill out a pre-determined suspected adverse drug reaction form once a side-effect is suspected. Moreover, the research assistant will be utilizing a suspected side-effect form and will be conducting an interview another day to assess the patient for any suspected side-effects.

Sample size

The sample size was estimated based on the anticipated difference (effect size) in the primary outcome between the two treatments (Tizanidine Vs Zolpidem) for the primary insomnia patients. The primary outcome considered was the mean global PSQI score before and after the treatment. We anticipated a medium effect size (Cohen's f = 0.25, Repeated measures ANOVA) for the primary outcome. The type I error alpha was set at 5%, and the power was set at 80%. The primary outcome will be measured four times (baseline, 4 weeks, 8 weeks, and 12 weeks), and the anticipated correlation among repeated outcome measures was 0.5. We also considered an attrition rate (dropout/lost follow up) of 10%. Therefore, the final sample size became 90 subjects (45 in each group). The calculation was done in G*Power version 3.1.9.7.

Data Analysis

Continuous variables will be presented as mean, median, standard deviation, and interquartile range, whereas categorical variables will be presented as frequency and percentage. Comparison of mean scores between two independent groups will be assessed using the independent samples t-test, whereas comparison of paired mean scores within the groups will be assessed using the paired samples t-test. A repeated measures ANOVA will be applied to evaluate the changes over time in the sleep quality between the two treatment groups. Association between two categorical variables will be assessed using a Chi-square test (Fisher's exact/Likelihood ratio). A P-value less than 0.05 will be considered statistically significant. All the analysis will be carried out in IBM SPSS Statistics (IBM Corp. Released 2022. IBM SPSS Statistics for Windows, Version 29.0. Armonk, NY: IBM Corp).

Ethical Considerations

Informed Consent:

In the informed consent process, all potential participants will receive detailed information about the study. A designated researcher from the study team will verbally explain the study in a language that is understandable to the participants. This discussion will take place in the outpatient sleep clinic and will be witnessed by another researcher to ensure transparency and accuracy. Any questions or concerns raised by the participants will be addressed at this time. Suppose the participant agrees to participate in the study. In that case, they will be provided with a comprehensive information and consent sheet outlining the study's purpose, procedures, potential risks and benefits, confidentiality measures, and their rights as participants. Subsequently, the participant will be asked to sign the consent form. Both the researcher who explained the study and the witnessing researcher will also sign the form to acknowledge the participant's informed consent.

Confidentiality:

All data collected throughout the study will be anonymized to remove any personally identifiable information. Additionally, measures will be implemented to ensure the secure storage of data. Access to study information will be restricted to authorized research personnel only, and data will be stored on a password-protected computer.

ELIGIBILITY:
Inclusion Criteria:

* Age and Gender Adult participants of either gender, aged 18-60 years old.
* Diagnosis: Diagnosed with primary insomnia by a psychiatry specialist, based on DSM-5 criteria.
* Consent: Able to provide written informed consent.
* Compliance: Willing to comply with study procedures and follow-up assessments.
* Medical Clearance: Participants must undergo a medical checkup by a medical officer affiliated with Al-Masarah Hospital before the randomization process. This checkup includes:
* Medical history review.
* Physical examination, including ECG.
* Vital signs check.
* Random blood sugar test.
* Laboratory evaluation (CBC, LFT, RFT, TFT, Lipid profile).
* Enrollment: Receiving medical clearance for enrollment in the study.

Exclusion Criteria:

* Secondary Insomnia: Individuals diagnosed with secondary insomnia.
* Substance Abuse History: Those with a history of substance abuse.
* Significant Medical or Psychiatric Disorders: Individuals diagnosed with significant and/or unstable medical or psychiatric disorders or mental retardation.
* Pregnancy or Lactation: Pregnant or lactating mothers, or those of childbearing potential not using an adequate method of contraception (excluding natural birth spacing methods).
* Drug Allergy: Known hypersensitivity or allergy to Tinazidine or Benzodiazepines.
* Communication Barriers: Individuals unable to understand or communicate with researchers.
* Recent Participation in Clinical Trials: Those who have participated in other clinical trials involving investigational drugs within the past 30 days before participation.
* Recent Use of Sleep Medication: Participants must not have taken any over-the-counter or prescription sleep medication within the past 30 days before participation.
* Use of Substances Affecting CNS: No intake of any substance with central nervous system (CNS) effects known to affect sleep within 30 days before participation.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Pittsburgh Sleep Quality Index | Baseline, 4 weeks, 8 weeks, 12 weeks
  Total Items: The PSQI contains a total of 24 questions. Range of Component Scores: Each component score ranges from 0 to 3 points. A score of 0 indicates no difficulty. A score of 3 indicates severe difficulty. Global PSQI Score: The seven component scores are summed to yield one "global" score.
  Range: The global score ranges from 0 to 21 points. A global score of 0 suggests no difficulty in any areas. A global score of 21 suggests severe difficulties in all areas.
  Interpretation of the Global Score:
  The global PSQI score is used to evaluate an individual's sleep quality. A global score greater than 5 often indicates significant sleep disturbances or poor sleep quality.

SECONDARY OUTCOMES:
Frequency and Severity of Side Effects | 4 weeks, 8 weeks, 12 weeks
  Documentation and assessment of the frequency and severity of side effects reported by patients using a self-report of suspected adverse drug reaction form.

IPD SHARING:
Plan to Share IPD: Yes